CLINICAL TRIAL: NCT01324947
Title: Open-label, Multi-center, Single Arm Study For The Safety And Efficacy Of Pomalidomide Monotherapy For Subjects With Refractory Or Relapsed And Refractory Multiple Myeloma. A Companion Study For Clinical Trial CC-4047-MM003
Brief Title: Study to Evaluate the Safety and Efficacy of Pomalidomide Monotherapy in Subjects With Refractory or Relapsed Refractory Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-MM-003/C; 2010-023343-16 (EudraCT Number)
Record Dates: First submitted 2011-03-27; First posted 2011-03-29 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; Relapsed Multiple Myeloma; Relapsed and Refractory Multiple Myeloma; Refractory Myeloma; Resistant Multiple Myeloma; Treatment-resistant Multiple Myeloma; Pomalidomide; Lenalidomide-resistant; Bortezomib-resistant; Companion
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Recurrence | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pomalidomide (Experimental): Oral pomalidomide 4 mg on Days 1-21 of 28-day cycle until progressive disease (PD) or unacceptable toxicity
  Interventions: Drug: pomalidomide

INTERVENTIONS:
Drug: pomalidomide — Oral pomalidomide 4 mg on Days 1-21 of 28-day cycle until progressive disease (PD) or unacceptable toxicity
  Other Names: CC-4047

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pomalidomide monotherapy in subjects with refractory or relapsed and refractory multiple myeloma who were enrolled in study CC-4047-MM-003 (NCT01311687) and discontinued treatment with high-dose dexamethasone due to disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with refractory or relapsed and refractory multiple myeloma who were enrolled in Study CC-4047-MM-003 and discontinued study therapy with dexamethasone alone (Treatment Arm B) after at least starting the second cycle of dexamethasone treatment and due to development of documented disease progression according to the International Myeloma Working Group (IMWG) criteria and as decided by an Independent Review Adjudication Committee (IRAC).
2. Must be ≥ 18 years at the time of signing the informed consent form.
3. The subject must understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted. The only exception is if a skeletal survey was performed within 90 days prior to the start of Cycle 1, then a new survey will not be required.
4. Must be able to adhere to the study visit schedule and other protocol requirements.
5. Subjects must have documented diagnosis of multiple myeloma and have measurable disease (serum M-protein ≥ 0.5g/dL or urine M-protein ≥ 200 mg/24 hours).
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
7. Females of childbearing potential (FCBP†) must agree to utilize two reliable forms of contraception simultaneously or practice true abstinence [when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception]from heterosexual contact for at least 28 days before starting study drug, while participating in the study (including dose interruptions), and for at least 28 days after study treatment discontinuation and must agree to regular pregnancy testing during this timeframe.
8. Females must agree to abstain from breastfeeding during study participation and 28 days after study discontinuation.
9. Males must agree to either use a latex condom during any sexual contact with FCBP or practice true abstinence [when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception] while participating in the study and for 28 days following discontinuation from this study, even if he has undergone a successful vasectomy. .
10. Males must also agree to refrain from donating semen or sperm while on pomalidomide and for 28 days after discontinuation from this study treatment.
11. All subjects must agree to refrain from donating blood while on study drug and for 28 days after discontinuation from this study treatment.
12. All subjects must agree not to share study medication

Exclusion Criteria

* The presence of any of the following will exclude a subject from enrollment:

  1. Subjects with multiple myeloma who were not treated as a part of Study CC-4047-MM-003 (Arm B).
  2. Subjects who received any anti-myeloma or anti-cancer therapies within the last 14 days of wash-out period before initiation of study treatment.
  3. Subjects who discontinued CC-4047-MM-003 study ≥120 days.
  4. Subjects who initiate another anti-myeloma therapy from the time of disease progression on study CC-4047-MM-003 to the time of treatment initiation in the companion study.
  5. Any of the following laboratory abnormalities:

     * Absolute neutrophil count (ANC) < 1,000/µL.
     * Platelet count < 75,000/µL for subjects in whom < 50% of bone marrow nucleated cells are plasma cells; or a platelet count < 30,000/µL for subjects in whom ≥ 50% of bone marrow nucleated cells are plasma cells
     * Creatinine Clearance < 45 mL/min according to Cockcroft-Gault formula (If creatinine clearance calculated from the 24-hour urine sample is ≥45 ml/min, patient will qualify for the trial)
     * Corrected serum calcium > 14 mg/dL (> 3.5 mmol/L);
     * Hemoglobin < 8 g/dL (< 4.9 mmol/L; prior RBC transfusion or recombinant human erythropoietin use is permitted)
     * Serum SGOT/AST or SGPT/ALT > 3.0 x upper limit of normal (ULN)
     * Serum total bilirubin > 2.0 mg/dL (34.2 μmol/L); or > 3.0 x ULN for subjects with hereditary benign hyperbilirubinaemia
  6. Prior history of malignancies, other than Multiple Myeloma (MM), unless the subject has been free of the disease for ≥ 5 years. Exceptions include the following:

     * Basal or Squamous cell carcinoma of the skin
     * Carcinoma in situ of the cervix or breast
     * Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)
  7. Hypersensitivity to thalidomide or lenalidomide. (This includes ≥ Grade 3 rash during prior thalidomide or lenalidomide therapy).
  8. Peripheral neuropathy ≥ Grade 2.
  9. Subjects who received an allogeneic bone marrow or allogeneic peripheral blood stem cell transplant less than 12 months prior to initiation of study treatment and who have not discontinued immunosuppressive treatment for at least 4 weeks prior to initiation of study treatment and are currently dependent on such treatment.
  10. Subjects who are planning for or who are eligible for stem cell transplant.
  11. Subjects with any one of the following:

      * Congestive heart failure (NY Heart Association Class III or IV)
      * Myocardial infarction within 12 months prior to starting study treatment
      * Unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris
  12. Subjects who received any of the following within the last 14 days of initiation of study treatment:

      * Plasmapheresis
      * Major surgery (kyphoplasty is not considered major surgery)
      * Radiation therapy
  13. Use of any investigational agents within 28 days or 5 half lives (whichever is longer) of treatment.
  14. Subjects with chronic conditions such as rheumatoid arthritis, multiple sclerosis and lupus, which likely need additional steroid or immunosuppressive treatments in addition to the study treatment.
  15. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
  16. Incidence of gastrointestinal disease that may significantly alter the absorption of pomalidomide.
  17. Subjects unable or unwilling to undergo antithrombotic prophylactic treatment.
  18. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
  19. Pregnant or breastfeeding females.
  20. Known human immunodeficiency virus (HIV) positivity or active infectious hepatitis A, B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2014-07-31 (Actual); Study Completion 2014-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Zaki, MD, PhD, Study Director — Celgene Corporation
Locations (91):
- Australia (9):
  - Royal Adelaide Hospital - SA Pathology Haematology, Adelaide
  - Princess Alexandra Hospital - Haematology, Brisbane
  - Royal Prince Alfred Hospital - Institute of Haematology, Camperdown
  - Peter McCallum Cancer Institute - Directorate of Cancer Medicine, East Melbourne
  - Frankston Hospital-Peninsula Health - Oncology Day Unit, Frankston
  - The Alfred Hospital - Malignant Haematology & Stem Cell Transplantation, Melbourne
  - Calvary Mater Newcastle - Haematology, Waratah
  - Border Medical Oncology, Wodonga
  - Wollongong Hospital - Haematology, Wollongong
- Belgium (3):
  - UZ Gent - Hematology, Ghent
  - University Hospital Leuven - Hematology, Leuven
  - Cliniques Universitaires ULC de Mont-Godinne - Hematology, Yvoir
- Canada (8):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver Centre, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Hospital, University Health Network, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
- Charles University Hospital - Internal Medicine, Prague, Czechia
- Denmark (4):
  - Aalborg Sygemus - Haematology, Aalborg
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense
  - Vejle Hospital - Hematology, Vejle
- France (13):
  - CHU Angers - Service des maladies du sang, Angers
  - Centre Hospitalier de la côte basque - Hematologie, Bayonne
  - Centre Hospitalier Départemental Vendée - Onco-hematologie, La Roche
  - CHRU de Lille - Service des maladies du sang, Lille
  - Institut Paoli Calmette - Hematology 1, Marseille
  - CHU Hôtel-Dieu - Hematologie, Nantes
  - Hôpital Saint Louis - Immuno-hematologie, Paris
  - CHU Saint Antoine - Service des maladies du sang, Paris
  - CHRU - Hôpital du Haut Lévêque - Centre François Magendie Service des maladies du sang, Pessac
  - Centre Hospitalier Lyon sud - Hematologie, Pierre-Bénite
  - CHRU Hôpital Purpan - Hematologie, Toulouse
  - Hôpital Bretonneau - Hématologie & Thérapie cellulaire, Tours
  - CHU Nancy - Hematologie, Vandœuvre-lès-Nancy
- Germany (10):
  - Universitatsklinikum Carl Gustav Carus-Medizinische Klinik und Poliklinik I, Dresden
  - Universitätsklinikum Essen, Klinik für Hämatologie Westdeutsches Tumorzentrum, Essen
  - Askepios Klinik Altona-Abteilung Hamatologie und Internistische Onkologie, Hamburg
  - Universitätsklinikum Heidelberg - Medizinische Klinik und Poliklinik V, Heidelberg
  - Universitätsklinikum Jena - Klinik fur Innere Medizin II-Hamatologie/Onkologie, Jena
  - Universitätsklinikum Leipzig - Medizinische Klinik und Poliklinik II, Leipzig
  - Universitätsklinikum Münster - Medizinische Klinik und Poliklinik A, Münster
  - Universitätsklinikum Tübingen - Medizinische Klinik und Poliklinik - Abteilung II, Tübingen
  - Universitätsklinikum Ulm - Klinik fur Innere Medizin III, Ulm
  - Universitätsklinikum Würzburg - Medizinische Klinik und Poliklinik II, Würzburg
- University of Athens - Alexandra Hospital, Athens, Greece
- Italy (9):
  - Università degli Studi di Bologna - Policlinico S. Orsola - Hematology, Bologna
  - AO Universitaria San Martino - hematooncology, Genova
  - Fondazione "G. Pascale" - Hematology, Napoli
  - Ospedale San Luigi AO Luigi Gonzaga - Hematology, Orbassano
  - Universita degli Studi di Padova - Clinical & Experimental Medicine, Padua
  - Ospedale Guglielmo da Saliceto - hematooncology, Piacenza
  - Unità di Ematologia Arcispedale S. Maria Nuova - Haematology, Reggio Emilia
  - Policlinico Umberto I, Università "La Sapienza" di Roma - Hematology, Roma
  - A.O.U. San Giovanni Battista - Hematology, Torino
- Netherlands (3):
  - VUMC - Hematology, Amsterdam
  - Erasmus Medical Center - Hematology, Rotterdam
  - University Medical Center - Hematology, Utrecht
- Russia (4):
  - Hematological Research Center under the Russian Academy of Medical Sciences - Hematology & BMT, Moscow
  - Moscow State Medical Institution Municipal Clinical Hospital n.a. S.P. Botkin - Hematology, Moscow
  - Russian Research Institute of Hematology and Blood Transfusion - Hematology, Saint Petersburg
  - State Higher Educational Institution St. Petersburg State Medical University - Onco-hematology, Saint Petersburg
- Spain (8):
  - Hospital Germans Trias i Pujol - Hematology, Badalona
  - Hospital Clinic i Provincial de Barcelona - Hematology, Barcelona
  - Hospital de Donostia - Hematology, Guipúzcoa
  - Hospital de La Princesa - Hematology, Madrid
  - Hospital 12 de Octubre - Hematology, Madrid
  - Hospital de Salamanca - Hematology, Salamanca
  - Hospital Universitario Marqués de Valdecilla - Hematology, Santander
  - Hospital La Fe - Hematology, Valencia
- Sweden (5):
  - Sahlgrenska Hospital, University of Goteborg - Hematology, Gothenburg
  - Karolinska University Hospital Huddinge - Center of hematology, Stockholm
  - Karolinska University Hospital-medicine, Stockholm
  - Karolinska University Hospital Solna- medicine, Stockholm
  - Overlakare Medocomcentrum - Hematology, Uppsala
- Switzerland (3):
  - Inselspital, Institut für Medizinische Onkologie, Bern
  - Hôpitaux Universitaire de Genève - Oncologie, Geneva
  - Klinik und Poliklinik für Onkologie - UniversitätsSpital Zürich, Zurich
- United Kingdom (10):
  - Royal Bournemouth Hospital - Haematology, Bournemouth
  - St James's University Hospital - Haematology, Leeds
  - St Bartholomew's Hospital - Medical Oncology, London
  - King's College Hospital - Haematology Clinical Trials, London
  - Freeman Hospital - Northern Centre for Cancer Care, Newcastle upon Tyne
  - Nottingham City Hospital - Centre for Clinical Haematology, Nottingham
  - Derriford Hospital - Haematology, Plymouth
  - Royal hallamshire Hospital - Haematology, Sheffield
  - Royal Marsden NHS Foundation Trust - Haematology, Surrey
  - Royal Wolverhampton Hospitals Trust - Research and Development, Wolverhampton

REFERENCES:
- [Background] Moreau P, Weisel KC, Song KW, Gibson CJ, Saunders O, Sternas LA, Hong K, Zaki MH, Dimopoulos MA. Relationship of response and survival in patients with relapsed and refractory multiple myeloma treated with pomalidomide plus low-dose dexamethasone in the MM-003 trial randomized phase III trial (NIMBUS). Leuk Lymphoma. 2016 Dec;57(12):2839-2847. doi: 10.1080/10428194.2016.1180685. Epub 2016 May 13. PMID 27173785
- [Background] Miguel JS, Weisel K, Moreau P, Lacy M, Song K, Delforge M, Karlin L, Goldschmidt H, Banos A, Oriol A, Alegre A, Chen C, Cavo M, Garderet L, Ivanova V, Martinez-Lopez J, Belch A, Palumbo A, Schey S, Sonneveld P, Yu X, Sternas L, Jacques C, Zaki M, Dimopoulos M. Pomalidomide plus low-dose dexamethasone versus high-dose dexamethasone alone for patients with relapsed and refractory multiple myeloma (MM-003): a randomised, open-label, phase 3 trial. Lancet Oncol. 2013 Oct;14(11):1055-1066. doi: 10.1016/S1470-2045(13)70380-2. Epub 2013 Sep 3. PMID 24007748
- [Background] Morgan G, Palumbo A, Dhanasiri S, Lee D, Weisel K, Facon T, Delforge M, Oriol A, Zaki M, Yu X, Sternas L, Jacques C, Akehurst R, Offner F, Dimopoulos MA. Overall survival of relapsed and refractory multiple myeloma patients after adjusting for crossover in the MM-003 trial for pomalidomide plus low-dose dexamethasone. Br J Haematol. 2015 Mar;168(6):820-3. doi: 10.1111/bjh.13227. Epub 2014 Nov 18. PMID 25403264

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: CC-4047-MM003C is a companion study for the trial CC-4047-MM-003 (NCT01311687). CC-4047-MM-003C enrolled those who discontinued treatment with dexamethasone alone (Treatment Arm B) in the CC-4047-MM-003 trial due to disease progression; those who had discontinued treatment with pomalidomide plus dexamethasone (Arm A) were not eligible to enroll
Groups:
- Pomalidomide: Oral pomalidomide 4 mg on Days 1-21 of each 28-day cycle until progressive disease (PD) or unacceptable toxicity
Period: Overall Study
Arm/Group | Pomalidomide
Started | 74
Safety Population | 73 (Safety Population includes those who were enrolled and received at least one dose of study drug)
Efficacy Evaluable Population (EEP) | 64 (Participants who received ≥ 1 dose of study drug and had at least 1 postbaseline efficacy assessment)
Completed | 0
Not Completed | 74
Not completed — Adverse Event | 7
Not completed — Death | 10
Not completed — Other | 3
Not completed — Progressive Disease | 50
Not completed — Withdrawal by Subject | 3
Not completed — 1 discontinued before starting drug | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was defined as all enrolled participants.
Arm/Group | Pomalidomide
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 42
Race [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 1
  Native Hawaiian or Other Pacific Islanders | 0
  White | 52
  Other | 2
  Not Collected | 19
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 49
  Not Collected | 19
Participants with Prior Anti-Myeloma (MM) Therapies [Number; unit: participants] | 74
Durie-Salmon Multiple Myeloma Stage before Study Entry [Number; unit: participants] — Stages are:
  Stage I: Hemoglobulin > 10 g/dL; serum calcium normal on roentgenogram; normal bone structure or solitary bone plasmacytoma only; Low M-component production rates (IgG value < 5 g/dL, IgA value < 3 g/dL; Bence Jones protein < 4 g/24h)
  Stage II: Overall data as minimally abnormal for stage I, and no single value as abnormal as defined for stage III
  Stage III: 1 or more of below:
  Hemoglobin < 8.5 g/dL; serum calcium > 12 mg/dL; Advanced lytic bone lesions (scale 3); High-M-component production rates (IgG value > 7 g/dL, IgA value > 5 g/dL; Bence Jones protein > 12 g/24h)
  participants
    Stage I | 8
    Stage II | 15
    Stage III | 50
    Missing | 1
Time From First Pathologic Diagnosis [Mean (Standard Deviation); unit: years] | 7.6 (3.72)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Objective Response According to International Myeloma Working Group (IMWG) Uniform Response Criteria Based on Investigator Assessment
Description: Objective response defined as a best overall response of stringent complete response (SCR), complete response (CR), very good partial response (VGPR) or partial response (PR) based on Investigator Assessment.
  SCR: CR and normal free light chain (FLC) ratio and no clonal cells in bone marrow; CR: Negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤5% plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein and urine M-protein level <100 mg/24 hours; PR: ≥50% reduction of serum M-Protein and reduction in urinary M-protein by ≥90% or to <200 mg/24 hours. A ≥50% decrease in the difference between involved and uninvolved FLC levels in place of the M-protein criteria or a ≥50% reduction in plasma cells in place of M-protein if baseline was ≥30%. If present at baseline a ≥50% reduction in size of soft tissue plasmacytomas.
Time Frame: From randomization through the study follow-up phase; up to the data cut-off of 31 July 2014; Maximum time on follow-up was 141.1 weeks.
Population: Intent to Treat Population was defined as all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Pomalidomide
Number analyzed (Participants) | 74
percentage of participants | 23.0

2. Secondary Outcome: Percentage of Participants With Objective Response According to European Group for Blood and Marrow Transplantation (EBMT) Criteria Based on Investigator Assessment
Description: Objective response defined as a best overall response of complete response (CR) or partial response (PR) based on the CR and requires all of the following:
  * Absence of original monoclonal paraprotein in serum and urine by immunofixation maintained at least 42 days.
  * <5% plasma cell in bone marrow aspirate and on bone marrow biopsy, if performed.
  * No increase in size or number of lytic bone lesions.
  * Disappearance of soft tissue plasmacytomas.
  PR requires all of the following:
  * ≥50% reduction in level of serum monoclonal paraprotein, maintained at least 42 days.
  * Reduction in 24-hour urinary light chain extraction by ≥90% or to <200 mg, maintained at least 42 days.
  * For patients with non-secretory myeloma, ≥50% reduction in plasma cells in bone marrow aspirate and on biopsy, if performed, for at least 42 days.
Time Frame: as for outcome 1
Population: Intent to treat population includes all participants enrolled.
Measure: Number; unit: percentage of participants
Groups:
- Pomalidomide: Oral pomalidomide 4 mg on Days 1-21 of 28-day cycle until progressive disease (PD) or unacceptable toxicity
  pomalidomide: Oral pomalidomide 4 mg on Days 1-21 of each 28-day cycle until progressive disease (PD) or unacceptable toxicity
Arm/Group | Pomalidomide
Number analyzed (Participants) | 74
percentage of participants | 20.3

3. Secondary Outcome: Number of Participants With Adverse Events and Type of Adverse Events
Description: An adverse event is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. A serious AE is any AE occurring at any dose that:
  * Results in death;
  * Is life-threatening;
  * Requires or prolongs existing inpatient hospitalization;
  * Results in persistent or significant disability/incapacity;
  * Is a congenital anomaly/birth defect;
  * Constitutes an important medical event.
  The Investigator assessed the relationship of each AE to study drug and graded the severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0):
  Grade 1 = Mild (no limitation in activity or intervention required); Grade 2 = Moderate (some limitation in activity; no/minimal medical intervention required);-Grade 3 = Severe (marked limitation in activity; medical intervention required, hospitalization possible); Grade 4 = Life-threatening; Grade 5 = Death
Time Frame: From first dose of study drug through to 30 days after the last dose, until the data cut-off date of 31 July 2014. Maximum time on treatment was 94.1 weeks.
Population: Safety population includes all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Pomalidomide
Number analyzed (Participants) | 73
participants
  Any adverse event | 73
  Grade 3-4 adverse event | 64
  AE related to pomalidomide | 51
  Grade 3-4 AE related to pomalidomide | 33
  Grade 5 AE | 19
  ≥1 Serious AE (SAE) | 52
  ≥1 SAE related to pomalidomide | 15
  ≥1 SAE leading to stopping pomalidomide | 6
  ≥AE leading to discontinuation of pomalidomide | 8
  ≥1 study drug related AE leading to stopping POM | 1
  ≥1 AE leading to reduction of pomalidomide | 11
  ≥1 study drug related AE leading to reducing POM | 9
  ≥1 AE leading to interruption of pomalidomide | 41
  ≥ 1 study drug related interruption of POM | 25

4. Secondary Outcome: Kaplan Meier Estimates for Progression Free Survival (PFS) by Investigator Based on IMWG
Description: Progression-free survival was calculated as the time from randomization to disease progression as determined by the Investigator based on the International Myeloma Working Group Uniform Response criteria (IMWG), or death on study, whichever occurred earlier.
  Progressive disease requires 1 of the following:
  * Increase of ≥ 25% from nadir in:
    * Serum M-component (absolute increase ≥ 0.5 g/dl)
    * Urine M-component (absolute increase ≥ 200 mg/24 hours)
    * In patients without measurable serum and urine M-protein levels the difference between involved and uninvolved free light chain (FLC) levels (absolute increase > 100 mg/dl)
    * Bone marrow plasma cell percentage (absolute % ≥ 10%)
  * Development of new or increase in the size of existing bone lesions or soft tissue plasmacytomas.
Time Frame: From randomization through the follow-up phase; Maximum duration of follow-up for PFS was 90.3 weeks.
Population: Intent to Treat included all participants enrolled.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide
Number analyzed (Participants) | 74
weeks | 16.0 [11.6 to 19.7]

5. Secondary Outcome: Kaplan-Meier Estimate for Time to Progression (TTP) Based on Investigator Assessment Using IMWG Criteria
Description: Time to progression (TTP) was calculated as the time from randomization to the first documented progression confirmed by the investigator and based on the International Myeloma Working Group Uniform Response criteria (IMWG).
  Progressive disease requires 1 of the following:
  * Increase of ≥ 25% from nadir in:
    * Serum M-component (absolute increase ≥ 0.5 g/dl)
    * Urine M-component (absolute increase ≥ 200 mg/24 hours)
    * In patients without measurable serum and urine M-protein levels the difference between involved and uninvolved free light chain (FLC) levels (absolute increase > 100 mg/dl)
    * Bone marrow plasma cell percentage (absolute % ≥ 10%)
  * Development of new or increase in the size of existing bone lesions or soft tissue plasmacytomas.
  * Development of hypercalcemia (corrected serum calcium > 11.5 mg/dl) attributed solely to plasma cell proliferative disease.
Time Frame: From randomization through the follow-up phase; up to the data-cut off of 31 July 2014; Maximum time to progression follow-up was 90.3 weeks.
Population: Intent to Treat includes all participants enrolled
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide
Number analyzed (Participants) | 74
weeks | 19.0 [14.1 to 27.4]

6. Secondary Outcome: Kaplan-Meier Estimate Duration of Response Based on Investigator Assessment Using IMWG Criteria
Description: Duration of Response (calculated for responders only) is defined as the time from the initial documented response (partial response or better) to confirmed disease progression by the investigator based on IMWG criteria.
Time Frame: From randomization through the study follow-up phase; up to the data cut-off of 31 July 2014; Maximum duration of response follow-up was 90.3 weeks.
Population: Includes those who had a partial response or better.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide
Number analyzed (Participants) | 17
weeks | 28.3 [8.1 to 53.4]

7. Secondary Outcome: Kaplan-Meier Estimate for Overall Survival
Description: Overall survival was calculated as the time from randomization to death from any cause. Overall survival was censored at the last date that the participant was known to be alive for participants who were alive at the time of analysis and for participants who were lost to follow-up before death was documented.
Time Frame: From randomization through the follow-up phase; Maximum time on follow-up was 141.1 weeks.
Population: Intent to Treat population included all participants enrolled into the study
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide
Number analyzed (Participants) | 74
weeks | 33.6 [26.4 to 66.3]

8. Secondary Outcome: Time to Response Based on IMWG and Assessed by the Investigator
Description: Time to Response was calculated as the time from enrollment to the initial response (PR or better) based on IMWG and assessed by the investigator.
Time Frame: From randomization through the follow-up phase; up to the data-cut off of 31 July 2014; Maximum time to response was 23.1 weeks
Population: Includes those who had at least a partial response or better; Intent to Treat
Measure: Median (Full Range); unit: weeks
Arm/Group | Pomalidomide
Number analyzed (Participants) | 17
weeks | 8.3 [4.1 to 23.1]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through to 30 days after the last dose, until the data cut-off date of 31 July 2014. Maximum time on treatment was 94.1 weeks.
Arm/Group | Pomalidomide
Serious Adverse Events (participants affected / at risk) | 52/73
Other Adverse Events (participants affected / at risk) | 68/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide (N=73)
Anaemia (Blood and lymphatic system disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Pneumonia (Infections and infestations) | 11
Bronchitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 2
Neutropenic sepsis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
General physical health deterioration (General disorders) | 8
Asthenia (General disorders) | 2
Pyrexia (General disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 2
Cachexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1
Hyperproteinaemia (Metabolism and nutrition disorders) | 1
Enterocolitis infectious (Infections and infestations) | 2
Septic shock (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Meningitis cryptococcal (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pneumonia streptococcal (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal infarction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Renal failure acute (Renal and urinary disorders) | 4
Renal failure (Renal and urinary disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Confusional state (Psychiatric disorders) | 2
Hip fracture (Injury, poisoning and procedural complications) | 1
Spinal cord compression (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide (N=73)
Anaemia (Blood and lymphatic system disorders) | 36
Neutropenia (Blood and lymphatic system disorders) | 35
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Leukopenia (Blood and lymphatic system disorders) | 9
Fatigue (General disorders) | 16
Pyrexia (General disorders) | 13
Asthenia (General disorders) | 7
Oedema peripheral (General disorders) | 6
Constipation (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Bronchitis (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 13
Hypercalcaemia (Metabolism and nutrition disorders) | 11
Decreased appetite (Metabolism and nutrition disorders) | 7
Headache (Nervous system disorders) | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Weight decreased (Investigations) | 6
Blood creatinine increased (Investigations) | 4
Insomnia (Psychiatric disorders) | 4
Renal failure (Renal and urinary disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may publish the results of its findings if a multicenter publication is not forthcoming within 18 months after study completion. Institution shall provide Celgene with a copy of the papers prior to submission; Celgene shall complete its review within 60 days after receipt. Upon Celgene's request, proposed publication or presentation will be delayed up to 60 additional days to enable Celgene to secure adequate intellectual property protection of patentable material.